CLINICAL TRIAL: NCT04671069
Title: A Single Center, Open-Label, Drug Interaction Study of MGL-3196 With Clopidogrel in Healthy Subjects
Brief Title: Drug Interaction Study of MGL-3196 With Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGL-3196-12
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Healthy
MeSH Terms: interventions — resmetirom; Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MGL-3196 100 mg tablet plus Clopidogrel 75 mg tablet (Experimental)
  Interventions: Drug: MGL-3196; Drug: Clopidogrel

INTERVENTIONS:
Drug: MGL-3196 — Administered orally on the morning of Day 1; Multiple-dose administration of 100 mg MGL-3196 on Day 6 until Day 14
Drug: Clopidogrel — After one-day washout period after Day 1, loading dose of 300 mg clopidogrel administered on Day 3 and then, at approximately the same time each morning, 75 mg clopidogrel administered on Days 4 to 11

SUMMARY:
The purpose of this study is to determine whether the single and multiple-dose pharmacokinetics (PK) of MGL-3196 are affected by co-administration with clopidogrel in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing and able to provide written informed consent
* Healthy, non-smoking male or female between the ages of 18 and 55 years (inclusive)
* Body weight > 50 kg and BMI between 18 and 32 kg/m2 (inclusive)
* Female subjects must:

  * Be non-pregnant and non-lactating
  * For females of non-childbearing potential, female must have undergone one of the following sterilization procedures at least 6 months prior to first dosing: hysterscopic fertilization bilateral salpingectomy, tubal occlusion, hysterectomy, bilateral oophorectomy
  * For postmenopausal women, are considered postmenopausal if amenorrheic for at least 12 months without an alternative medical cause
  * For females of childbearing potential, must one of the following birth control methods: surgical sterilization of partner, hormonal contraceptives no prone to drug-drug interactions, hormonal oral contraceptive agents such as normal and low dose combined pills or progesterone only pills, physical barrier method (eg, male condom) in addition to spermicide, non-hormonal intrauterine device for at least 3 months prior to first dosing, total abstinence from sexual intercourse for at least 3 months prior to first dosing and through study completion
* If male and non-vasectomized, must agree to use a condom with spermicide or abstain from sexual intercourse from the first dose of study drug until 14 days beyond the last dose of study drug. No restrictions required for vasectomized male provided his vasectomy has been performed 3 months or more prior to Day 1. A male who has been vasectomized less than 3 months prior to study start must follow the same procedure as a non-vasectomized male.

Exclusion Criteria:

* Any clinically significant abnormal findings on physical examination, clinical laboratory tests or 12-lead ECG.
* Evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, renal, hepatic, neurological or psychiatric disease.
* Current or recent (< 6 months) hepatobiliary disease; or AST, ALT or direct bilirubin greater than the upper limit of reference range at screening. Repeat testing is allowed per site standard procedures.
* Gilbert's syndrome.
* Pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of study drug (Cholecystectomy is allowed).
* Abnormal screening ECG: including machine-read QTcF >450 msec in men and QTcF > 470 msec in women (confirmed by manual over read) or any rhythm other than normal sinus rhythm which is interpreted by the Investigator to be clinically significant.
* History of sensitivity to a similar study drug, thyroid medication, or a history of important drug or other allergy (except for untreated, asymptomatic seasonal allergies at time of dosing) unless deemed not clinically significant by the Investigator.
* Participation in another clinical trial of an investigational drug (or medical device) within the last 30 days prior to the Day 1, or who have been exposed to more than four new chemical entities within 12 months prior to Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-14 (Actual)

PRIMARY OUTCOMES:
AUC from the time of dosing of clopidogrel as affected by single and multiple daily dosing with MGL-3196 100 mg/day in healthy subjects | 14 days
Pharmacokinetics (Cmax) of clopidogrel as affected by chronic dosing with MGL-3196 100 mg/day in healthy subjects | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No